CLINICAL TRIAL: NCT02043964
Title: Tear Analysis by Isoelectric Focusing in Clinically Isolated Syndrome as Multiple Sclerosis Criterion Among Patients With or Without Lesions at the Magnetic Resonance Imaging (Oligoclonal Profile of Tears)
Brief Title: Tear Analysis by Isoelectric Focusing in Clinically Isolated Syndrome as Multiple Sclerosis Criterion
Acronym: POLAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lille Catholic University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RC-P0021
Record Dates: First submitted 2013-11-22; First posted 2014-01-23 (Estimated); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: Clinically Isolated Syndrome; Multiple Sclerosis
Keywords: Multiple Sclerosis; Clinically Isolated Syndrome; Tears; Isoelectric focusing; Oligoclonal profile
MeSH Terms: conditions — Multiple Sclerosis; Lacerations

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- tears and cerebro-spinal fluid sampling (Experimental)
  Interventions: Procedure: tears and cerebrospinal fluid sampling

INTERVENTIONS:
Procedure: tears and cerebrospinal fluid sampling — All patients recruited in this study will undergo a cerebrospinal fluid sampling which is an invasive procedure included in the actual routine practice. In addition a sampling from eyes will be obtain using the Schirmer test to get tears from the lacrimal gland.

SUMMARY:
This is a multicentric and prospective study for the validation of a diagnostic method in multiple sclerosis. Our hypothesis is that there is a characteristic profile of tears that can be recognized in order to help in the diagnosis of this pathology and that could possibly replace the lumbar punction which is an invasive method. Semi-automatic and automatic techniques of isoelectric focusing will be developed for analyzing data from tears. These results will help in the identification of markers of this disease.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old or more
* Clinically isolated syndrome of less than 3 months of onset
* Informed consent to participate

Exclusion Criteria:

* Progressive primary multiple sclerosis
* Relapsing remitting multiple sclerosis
* Persons wearing contact lenses
* Ocular Infection
* Corticoid treatment at least 30 days before sampling
* Immunosuppressive or immunomodulatory treatment at least 3 months before sampling
* Pregnancy or breast feeding
* No coverage by the Social Insurance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 165 (Actual)
Dates: Start 2012-10; Primary Completion 2018-06 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Test of the concordance coefficient between the analysis of tears and the analysis of cerebrospinal fluid | two years after
  Test of the concordance coefficient between the analysis of tears and the analysis of cerebrospinal fluid

SECONDARY OUTCOMES:
Diagnostic performance of isoelectric focusing of tears | inclusion, two years after
  Identification of the number of patients with a typical electrophoretic profile in tears allowing the early diagnosis of a SEP-RR
Concordance between visual and automatic reading of electrophoretic profiles | two years
  Determination of percentage of positive and negative tests after visual and automatic reading of electrophoretic profiles
Calculation of sensitivity/specificity | two years
  Calculation of sensitivity/specificity
Calculation of positive/negative predictive value | two years
  Calculation of positive/negative predictive value
Calculation of efficiency odds ratio | two years
  Calculation of efficiency odds ratio

CONTACTS AND LOCATIONS:
Overall Officials: Gérard Forzy, MD, Study Director — Groupement des Hôpitaux de l'Institut Catholique de Lille; Patrick Hautecoeur, MD, Principal Investigator — Groupement des Hôpitaux de l'Institut Catholique de Lille; Patrick Vermersch, MD, PhD, Principal Investigator — Centre Hospitalier Régional, Universitaire de Lille; Gilles Defer, MD, Principal Investigator — Centre Hospitalier Universitaire Caen; Christine Lebrun-Fresnay, MD, PhD, Principal Investigator — Centre Hospitalier Universitaire de Nice; Jérôme de Seze, MD, PhD, Principal Investigator — Centre Hospitalier Régional Universitaire de Strasbourg; Thibault Moreau, MD, Principal Investigator — Centre Hospitalier Universitaire Dijon; Pierre Clavelou, MD, Principal Investigator — University Hospital, Clermont-Ferrand; Olivier Heinzlef, MD, Principal Investigator — Centre Hospitalier Intercommunal Poissy-St-Germain; Christian Confavreux, MD, Principal Investigator — Centre Hospitalier Universitaire de Lyon; Marc Debouverie, MD, PhD, Principal Investigator — Central Hospital, Nancy, France; Jean Pelletier, MD, PhD, Principal Investigator — Hopital de la Timone, Marseille; Bruno Brochet, MD, PhD, Principal Investigator — University Hospital, Bordeaux; Sandrine Wiertlewski, MD, Principal Investigator — Nantes University Hospital; Albert Verier, MD, Principal Investigator — Centre Hospitalier de Valenciennes; Bertrand Bourre, MD, Principal Investigator — University Hospital, Rouen
Locations (15):
- France (15):
  - Centre Hospitalier Universitaire de Bordeaux, Bordeaux
  - Centre Hospitalier Universitaire Caen, Caen
  - Centre Hospitalier Universitaire de Clermont-Ferrand, Clermont-Ferrand
  - Centre Hospitalier Universitaire de Dijon, Dijon
  - Centre Hospitalier Régional Universitaire de Lille, Lille
  - Groupe Hospitalier de l'Institut Catholique de Lille, Lomme
  - Centre Hospitalier Universitaire de Lyon, Lyon
  - Hopital de la Timone, Marseille
  - Universitaire de Nancy, Nancy
  - Centre Hospitalier Universitaire de Nantes, Nantes
  - Centre Hospitalier Universitaire de Nice, Nice
  - Centre Hospitalier Intercommunal Poissy-St-Germain, Poissy
  - Centre Hospitalier Univetrsitaire de Rouen, Rouen
  - Centre Hospitalier Régional Universitaire de Strasbourg, Strasbourg
  - Centre Hospitalier de Valenciennes, Valenciennes